CLINICAL TRIAL: NCT03047902
Title: Disclosure of Smoking in Adolescents With Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: The Whittington Hospital NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202314
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Adolescent Smoking Cessation Asthma Carbon Monoxide.
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent Present (Active Comparator): The adolescents in group 1 (Parent Present) will be aware that their parents will be able to share the information on the questionnaire, but they will be assured of the confidentiality of the CO test. This will also be explained to the parent.
  Intervention: Parents will be present for the questionnaire but not for the CO test.
  Interventions: Other: Group 1 - Parents will be present for the Questionnaire.
- Parent Absent (Active Comparator): The adolescents in group 2 (parents not present) will be assured of the confidentiality of the questionnaire and CO test. The confidentiality of the test will also be explained to the parent.
  Intervention: Parents will not be present for the questionnaire or the CO test
  Interventions: Other: Group 2- Parents will not be present for the Questionnaire

INTERVENTIONS:
Other: Group 1 - Parents will be present for the Questionnaire. — In Group 1 the parents will be present for the questionnaire. The information on the questionnaire will be disclosed to them.
  In Group 2 the parents will not be present for the questionnaire and the information will not be disclosed to them.
  Arms: Parent Present
Other: Group 2- Parents will not be present for the Questionnaire
  Arms: Parent Absent

SUMMARY:
This is an exploratory randomised matched cohort pilot study. It is hypothesised that adolescents (aged 13-16 years) with asthma attending a secondary care outpatient asthma clinic, will disclose their smoking status to a doctor or nurse, if questioned alone without a parent present and if advised that they will have biological validation of their smoking status using a carbon monoxide monitor. It is a study of 30 subjects, who will be recruited over a period of 6 months.

DETAILED DESCRIPTION:
Background:

There are currently no recommendations for how to obtain accurate information on tobacco use from teenagers aged 13-16 years, who have asthma and are attending a secondary care outpatient clinic. The approach adopted in this study, using a simple questionnaire and Carbon Monoxide monitor to verify smoking status, could potentially allow health care professionals to identify at risk adolescents before they become regular smokers. It is proposed that adolescents will disclose more accurate information about their smoking status if questioned alone without a parent present and if advised that they will have biological validation of their smoking status, using a carbon monoxide monitor.

The objectives of the study are:

1. Use a smoking questionnaire, which will be designed with patient and parent feedback and contribution, to measure smoking status in adolescents, attending a secondary care outpatient clinic.
2. To assess the appropriateness and acceptability of Carbon Monoxide(CO) monitoring to correlate smoking status in adolescents attending a paediatric outpatient clinic.

Design and Methodology:

All patients will be selected from the paediatric asthma clinic list at Whittington Health. The researcher will approach them with information regarding the research using a Participant Information Sheet. The CO test and the interpretation of the results of the CO test will be explained also. The researcher will consent both the parents and adolescents in both groups for the study and CO test. The adolescent will need to give written informed consent. The adolescents in group 1 (parents present) will be aware that their parents will be able to share the information on the questionnaire, but they will assured of the confidentiality of the CO test. This will also be explained to the parent. The adolescents in group 2 (i.e. parents present) will be assured of the confidentiality of the questionnaire and CO test. The confidentiality of the results will also, be explained to the parent. The parents will consent for their child to take part in the study but the teenagers will also be asked to assent to the study. It would be made clear to the parent that the teenager has a choice to participate and their refusal is not necessarily related to the fact that they may smoke. Irrespective of whether they participate or not all parents and teenagers will have smoking advice discussed with them.

Each consenting participant will be given a short questionnaire to complete. This will include 5-6 questions about their smoking history and how much they smoke and if they have ever tried to give up and how. The questionnaire will also request some basic demographic data and postcode to help identify the potential effects of environmental pollution and passive smoking may have on the results. The questionnaire should take no longer than 5 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 13-16 years of age at the time of the study.
* Participants will be regular patients of the asthma clinic and will have a diagnosis of asthma
* All patients will have a consultant verification of their asthma diagnosis
* Patients with multisystem atopy will be included in the study
* Only patients accompanied by parents and with parental consent will be enrolled to the study.

Exclusion Criteria:

* Patients <13 years
* Patients attending clinic without a parent.
* Patients with special educational needs or communication difficulties
* Patients who don't speak English as a first language, if an interpreter is not

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Ascertaining smoking status in adolescents with asthma. | 6 months
  To ascertain if adolescents with asthma are more likely to be truthful about smoking status if questioned alone without their parents and with knowledge that this will be verified by carbon monoxide monitoring. This may provide scope for a personal intervention approach to facilitate discussion about smoking cessation intervention strategies and also may be able to be extrapolated to all paediatric outpatient units and GP surgeries.

SECONDARY OUTCOMES:
Evidence base for protocol/guidance | 1 year
  To provide an evidence base for producing a guidance/protocol for how best to obtain a smoking history from adolescents in a collaborative and facilitative way.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Hakim, PHD, Principal Investigator — Imperial College London
Locations (1):
- Whittington Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No